CLINICAL TRIAL: NCT00493597
Title: Blood Endothelium Progenitor Cells and Dendritic Cells as Novel Predictive Biomarkers of In-stent Restenosis After Percutaneous Coronary Intervention.
Brief Title: Blood Endothelium Progenitor Cells and Dendritic Cells as Predictive Biomarkers of In-stent Restenosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Steven Haine, Dr.S.Haine, University Hospital, Antwerp
Other Study IDs: EC 7/5/36
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Atherosclerosis; Restenosis
Keywords: Atherosclerosis; Restenosis; EPC; DC
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
clinically relevant in stent restenosis occurs in 5-10% of the non-diabetic patients treated with a coronary bare metal stent. Recent research has identified endothelial progenitor cells as well as dendritic cells as components of neointima. Numerical and functional evaluation of endothelial progenitor and dendritic cells at the time of coronary stent implantation is assessed and the relation with clinical and/or angiographic restenosis at 6 months post-stent implantation is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* Scheduled for PCI
* Candidate for CABG if necessary
* Clinical evidence of ischemic heart disease and/or abnormal functional study
* New native coronary artery lesion >50%-<100% stenosis
* Lesion length<30 mm, treatment with a single bare metal stent planned
* Reference diameter 2.5-3.5 mm
* Informed consent explained, red, understood and signed by the patient

Exclusion Criteria:

* Pregnancy, birth or lactation period <6 months ago
* Women of childbearing age who do not intend to use accepted anticonceptive measures or who wish to get pregnant
* Left ventricular ejection fraction <30%
* Acute myocardial infarction (ST-elevation, Q-wave evolution or CK-MB >2x upper limit of normal)in the past month
* Contra-indication to PCI
* Diabetes mellitus
* Planned drug eluting stent implantation
* Total occlusion (TIMI 0 or 1)
* Ostial localisation (<3.0 mm of the coronary ostium) of the lesion
* Bifurcational lesion with side branch >2.0 mm or side branch which will be recanalised at occlusion due to PCI
* Lesion in arterial or venous bypass or anastomosis with coronary
* Angiographic contra-indication to IVUS
* Severe renal insufficiency (creatinine clearance <30 mL/')
* Severe hepatic insufficiency
* Systemic inflammatory pathology of any kind
* Uncorrected hyperthyreosis
* Hematologic or other malignancy, prior radio- or chemotherapy
* Severe peripheral artery disease (accesproblem via groin)
* Use of corticosteroïds or immune suppression therapy
* Contrastallergy
* Life expectancy <1 year
* Participation in other clinical study which has not ended yet

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-diabetic patients scheduled for PCI with a single bare metal stent in a significant de novo coronary lesion
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2007-10; Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Haine, MD, Principal Investigator — UZ Antwerpen
Locations (1):
- Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen, Belgium